CLINICAL TRIAL: NCT02755285
Title: A Concurrence Study of Diagnostic Visualization Comparing Blue Light Imaging (BLI) With Flexible Spectral-Imaging Color Enhancement (FICE)
Brief Title: Study Comparing Blue Light Imaging (BLI) With Flexible Spectral-Imaging Color Enhancement (FICE)
Acronym: BLI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-16-004
Record Dates: First submitted 2016-04-13; First posted 2016-04-28 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Endoscopy
Keywords: BLI; FICE
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Endoscopy Procedure (Experimental): All subjects will have 1 endoscopy procedure, in which they will have a white light examination followed by FICE and BLI imaging on a maximum of two (2) anatomical sites per subject.
  Interventions: Device: Single Endoscopy Procedure

INTERVENTIONS:
Device: Single Endoscopy Procedure — All subjects will have 1 endoscopy procedure, in which they will have a white light examination followed by FICE and BLI imaging on a maximum of two (2) anatomical sites per subject.

SUMMARY:
The study is intended to demonstrate substantial equivalence of visualization using BLI to the predicate device, FICE, so as to support the addition of BLI as an adjunct to white light imaging in the company's video processor.

DETAILED DESCRIPTION:
This clinical study will consist of acquisition of images, followed by a reader study.

ELIGIBILITY:
Inclusion Criteria:

* Referred for clinically indicated gastrointestinal diagnostic endoscopy
* Ability to understand the requirements of the study, to provide written informed consent and to comply with the study protocol
* Ability to understand and provide written authorization for the use and disclosure of protected health information (PHI) per the Health Insurance Portability and Accountability Act (HIPAA) privacy ruling.

Exclusion Criteria:

* Under the age of 21 years
* Is an inmate (see US Code of Federal Regulations 45 C.F.R. 46.306)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aiji Matsunuma, Study Director — FUJIFILM Medical Systems, U.S.A., Inc.
Locations (1):
- Mayo Clinic AZ, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled had been referred to Mayo Clinic for clinically indicated gastrointestinal diagnostic endoscopy between August 19, 2016 and September 7, 2016.
Pre-assignment Details: Each subject underwent a complete diagnostic endoscopy examination with white light, followed by an exam with BLI (BLI + BLI-brt) and FICE, at 3 FICE settings (1,2 & 6). Each subject could contribute up to 2 anatomical sites (regions of interest).
Period: Overall Study
Arm/Group | Single Endoscopy Procedure
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Endoscopy Procedure
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 58.6 [39 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Image Quality Scores Using Likert Scale
Description: Likert score ratings of image quality for Blue Light Imaging (BLI), Blue Light Imaging-bright (BLI-brt) and Flexible spectral-Imaging Color Enhancement (FICE) images. Each BLI and BLI-Brt setting was compared to FICE, to determine which settings were equivalent to FICE.
  Likert Score Scale:
  1. Not seen;
  2. poor but usable, characteristic features are detectable but details are not fully reproduced; features just visible;
  3. good; allows an adequate assessment, details of anatomical structures are visible but not necessarily clearly defined; details emerging;
  4. very good; allows an excellent assessment, anatomical details are clearly defined; details clear
  This was a blinded and randomized Reader assessment of all BLI and FICE images.
Time Frame: Two to three months
Population: All patients had imaging done with white light (standard) as well as BLI, BLI-brt, and FICE. Each of the three (3) Readers had a unique set of randomized images which they reviewed independently during the reader study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Endoscopy Procedure
Number analyzed (Participants) | 20
units on a scale
  BLI | 3.3 (0.2)
  BLI-brt | 3.5 (0.1)
  FICE Setting 1 | 3.4 (0.1)
  FICE Setting 2 | 3.5 (0.1)
  FICE Setting 6 | 3.5 (0.0)

ADVERSE EVENTS:
Arm/Group | Single Endoscopy Procedure
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No